CLINICAL TRIAL: NCT00948727
Title: Reduction of Acute and Chronic Graft-versus-host Disease After Allogeneic Hematopoietic Stem-cell Transplantation by Adapting Cyclosporine Doses According to Calcineurin Activity : a Proof-of-concept Trial
Brief Title: Cyclosporine Dose Adjustment According to Calcineurin Activity After Allogeneic Hematopoietic Stem-cell Transplantation
Acronym: CALCICLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Thérèse NGOUE, Department Clinical Research of developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P021004
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-07

CONDITIONS: Hematopoietic Stem Cell Transplantation; Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose adjustment according CN activity (Experimental)
  Interventions: Behavioral: Dose adaptation according to CN activity monitoring; Drug: Cyclosporine (CsA)

INTERVENTIONS:
Behavioral: Dose adaptation according to CN activity monitoring — The protocol of the CALCICLO trial consisted in a CsA dose adaptation during the first 100 days following transplantation. This dose adaptation was performed according to both residual CsA blood and CN activity levels only if the safety of vital functions - especially renal, liver, and neurological - was preserved as assessed by clinical evaluations and laboratory analyses such as creatinine clearance higher than 40 ml/min, serum bilirubin lower than 40 µM and absence of neurological signs. According to the protocol, CsA blood levels and CN activity were measured concomitantly at least once a week from day 0 to day 15, twice a week from day 16 to day 35 and then once a week until day 100.
Drug: Cyclosporine (CsA) — Cyclosporine (CsA)

SUMMARY:
The purpose of this trial is to assess whether an adaptation of cyclosporine (CsA) dose according to a longitudinal calcineurin (CN) activity monitoring would prevent the onset of graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
Our previous studies established a correlation between increased calcineurin (CN) activity and the risk of developing severe acute GVHD in allogeneic stem cell transplant recipients receiving immunosuppressive therapy with calcineurin inhibitors.

This proof-of-concept trial is aiming at evaluating CALCIneurin activity as a monitoring biomarker of efficacy of cyCLOsporine - (CALCICLO) - for the prophylaxis of acute GVHD. Our aim is to assess whether a longitudinal monitoring of CN activity would permit to adapt and optimize the dose of CsA that would prevent the onset of severe acute GVHD, yet still maintaining an acceptable tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients were between the age of 12 and 60 years
* Patients planned to receive an allogeneic HSCT following a myeloablative conditioning regimen

Exclusion Criteria:

* Transplant from a syngeneic donor
* Evidence of refractory disease
* Nonmyeloablative conditioning
* Any participation to a study with a new investigational drug within the previous 3 months

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-01; Primary Completion 2006-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary end point is the acute grade II to IV GVHD-free survival 100 days after transplantation. | 100 days after transplantation.

SECONDARY OUTCOMES:
Safety was a secondary endpoint. It was assessed through clinical assessments including vital signs, creatinine clearance, the presence or not of neurological signs evocative of, or consistent with CsA toxicity, creatinine clearance and serum bilirubin. | 100 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Sanquer, Pharm.D., Study Director — AP-HP, Hôpital Necker-Enfants Malades
Locations (1):
- Chu Henri Mondor, Créteil, France

REFERENCES:
- [Background] Sanquer S, Schwarzinger M, Maury S, Yakouben K, Rafi H, Pautas C, Kuentz M, Barouki R, Cordonnier C. Calcineurin activity as a functional index of immunosuppression after allogeneic stem-cell transplantation. Transplantation. 2004 Mar 27;77(6):854-8. doi: 10.1097/01.tp.0000114612.55925.22. PMID 15077026